CLINICAL TRIAL: NCT04085861
Title: Mental Health in Dancers; an Intervention Study
Acronym: MeHeDa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Norwegian association for youth mental health (Unknown); Østfold University College (Unknown)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19/00770
Record Dates: First submitted 2019-09-06; First posted 2019-09-11 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Mental Health Impairment; Mental Health; Eating Disorders; Perfectionism; Depression, Anxiety; Coping Behavior; Self Esteem; Body Image; Body Weight
Keywords: Mental health; Eating disorders; Perfectionism; Body image; Body dissatisfaction; Body appreciation; Depression; Energy availability
MeSH Terms: conditions — Psychological Well-Being; Feeding and Eating Disorders; Depression; Anxiety Disorders; Body Weight

STUDY DESIGN:
Intervention Model Description: Professional dancers at the Norwegian University of Dance (NDH) (n=200) and a group of control persons (Oslo National Academy of the Arts) (n=100) are asked to take part in this study. NDH students receive an intervention after pre-tests and are re-evaluated post-intervention and 6 months post-intervention. The art students responds to similar questionnaires at the three evaluation times. Additionally, the dance teachers (n=50) are evaluated pre, post and 6-months post-intervention, receiving a specific intervention designed for teachers on mental health literacy and which actions to take if findings dancers with mental health issues.
Who Masked: Outcomes Assessor
Masking Description: By using id-numbers for each respondent in this trial, the outcome assessor will not be able to identify the group of responders.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dancers (Experimental): Recruited group of professional dancers from the Norwegian University of dance
  Interventions: Behavioral: Mental health literacy in dancers
- Control (No Intervention): Recruited group of professional art students from the Oslo Academy of the Arts (Norway)
- Dance teachers (Experimental): Recruited group of dance teachers from the Norwegian University of dance
  Interventions: Behavioral: Mental health literacy in dance teachers

INTERVENTIONS:
Behavioral: Mental health literacy in dancers — Receive a designed informative intervention (3 workshops of 90min each) aimed at improving their knowledge and skills on proper recovery, performance nutrition, and mental health literacy.
  Arms: Dancers
Behavioral: Mental health literacy in dance teachers — Receive a designed informative intervention (3 workshops of 60min each) aimed at improving their knowledge and skills on how to identify and deal with mental health- and nutritional issues in dancers.
  Arms: Dance teachers

SUMMARY:
International studies reveal high prevalence of eating disorders (ED) and mental health issues amongst professional dancers, and the Norwegian National Ballet's house previously (2005) reported a lifetime prevalence of ED by 50% amongst female ballet dancers. Mental health issues and ED have been acknowledged for several years in most sports; still the same do not apply to dance sports. The objective of this study is to improve the knowledge on prevalence of mental health issues in professional dancers and the corresponding awareness of such among dance teachers. Additional objectives are to evaluate the effect of an intervention aimed to improve knowledge on nutrition, recovery strategies and mental health literacy among professional dancers and their teachers.

DETAILED DESCRIPTION:
It is well documented that professional dancing increases the risk for, or strongly associates to, mental health issues like eating disorders, anxiety, and compulsive-obsessive disorders. As much as the international sport society has acknowledged the challenges on ED in sport, the same do not apply to dance. The point prevalence of ED in the general european population is about 0.3-4.0%, with a corresponding prevalence amongst professional dancers of 12.0-26.5%. Furthermore, the highest risk for ED among dance discipline is found to be within ballet. There are no reports on prevalence in Norwegian dancers; however, the Norwegian National Ballet's house reports a lifetime prevalence of 50% amongst ballet dancers. Previous studies have identified low knowledge and practice on performance nutrition and weight regulation strategies among dancers and their teachers. Findings indicates high risk of low energy availability, implying a high risk for the many associated negative effects on physical and mental health and performance capacity. Additionally, studies finds high levels of body dissatisfaction, body weight concern, perfectionism and low self-esteem, and also high prevalence of anxiety and depression.

Several intervention studies finds positive effect on body dissatisfaction, disordered eating behaviour, nutritional intake in sport athletes, and also in ballet dancers in the US and Canada. Nevertheless, so far there haven't been any intervention in Norwegian dancers.

The objective with this study is to explore mental health in professional dancers and their knowledge on recovery strategies and nutritional needs, and to implement and evaluate the effect of an intervention designed to improve these aspects. A group of performance art students serves as control to the intervention effect. Additionally this study evaluates the knowledge of these issues amongst dancers and how to deal with such issues, in dance teachers, and aims to implement and evaluate the effect of an intervention designed to improve the knowledge on these aspects.

ELIGIBILITY:
Inclusion Criteria:

* professional dancers at the Norwegian University of dance
* dance teacher at the Norwegian University of dance
* art student at the Oslo National Acadmey of the Arts

Exclusion Criteria:

* Not student or dance teacher at the Norwegian University of dance, or student at the Oslo National Acadmey of the Arts

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of eating disorders | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Eating disorder examination questionnaire (EDE-q) by Prof. Fairburn validly assesses the frequency and severity of ED features to produce ED diagnoses according to the DSM-5. It constitutes 22 items scored on a Likert scale from 0-6 and 6 items in which a number of frequency is given for a given eating behavior. The questionnaire is averaged with a global scale and 4 subscales, in which a higher value indicates higher clinical severity. The global score cut-off score indicating probability of an eating disorder in the Norwegian female population is 2.5.

SECONDARY OUTCOMES:
Change in perfectionism | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Children and adolescent perfectionism scale (CAPS) is a 22-item measure of perfectionism in children and adolescents, compromising two subscales; self-oriented perfectionism (12 items) and social-oriented perfectionism (10 items). Questions rates from 1 (false - not at all true) to 5 (very true for me); hence a higher value indicates higher level of perfectionism.
Change in resilience | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Resilience scale for adults (RSA) can be used to assess the presence of protective factors important to regain and maintain mental health. It is a self-report instrument for evaluating six protective dimensions of resilience in adults: (1) Perception of the Self, (2) Planned Future, (3) Social Competence, (4) Family Cohesion, (5) Social Resources, (6) Structured Style. The RSA has 33 items; item-response ranges from one to seven; higher scores reflect higher levels of protective factors of resilience.
Change in self esteem | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Rosenborg Self esteem inventory by Rosenberg, M. (1965). A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The scale is believed to be uni-dimensional. All items are answered using a 4-point Likert scale format ranging from strongly agree to strongly disagree.
Change in body appreciation | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Body appreciation scale (BAS-2) by Avalos et al 2005. The 10-item Body Appreciation Scale ) assesses individuals' acceptance of, favorable opinions toward, and respect for their body. Each item is scored on a Likert scale from 1-5, and global score is the average score for items 1-10.
Change in energy availability | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Low energy availability in females questionnaire (LEAF) and Low energy availability in males questionnaire (LEAM). The LEAF-Q was developed to screen for LEA in female athletes, and measures occurrence of injuries, gastrointestinal dysfunction (GD) and menstrual irregularities (MI) related to low energy availability. Suggested cut-off's's for GD, MI, and for the total LEAF-Q score are ≥2, ≥4, and ≥8, respectively, with higher scoring indicating more severe clinical condition. The LEAM-q is a male-adapted version of the questionnaire, which is currently under validation.
Change in depression and anxiety | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Hopkins symptom check list (SCL-10) is used to measure psychological distress among adolescents and adults; designed to measure the symptoms of anxiety and depression. Four of the ten questions are about anxiety and six are about depression. All 10 questions have 4 response categories: 'Not at all', 'A little', 'Quite a bit' and 'Extremely'. The responses are summarized across all items and the mean score is used as a measure of psychological distress. An average score ≥1.85 is considered a valid cut-off value for prediction of mental distress.

OTHER OUTCOMES:
Change in demographic information | Pre-intervention, post-intervention (4-months), and follow up (6-months post-intervention)
  Age, body weight, height, history with sports, knowledge on nutrition, knowledge on recovery strategies
Personal experiences | Pre- and post-intervention (4-months)
  Individual interviews with dancers and dance teachers on their knowledge and experiences with mental health as a dancer/within dancers, and with their sport and its measures in providing optimal physical and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Beate Anstensrud, MSc, Study Director — Norwegian association for youth mental health
Locations (1):
- Norwegian School of Sports Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Results from study belongs to the persons and institutions behind this study